CLINICAL TRIAL: NCT05058859
Title: Long Term Clinical Efficacy of Sodium-glucose Cotransporter-2 (SGLT-2) Inhibitor in Cystinurics
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was never secured so clinical trial was never started; this study was abandoned
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGLT2 1 Year
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Cystinuria
MeSH Terms: conditions — Cystinuria | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Drug (Experimental): The study drug is Dapagliflozin
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin is to lower blood sugar levels in adults with type 2 diabetes
  Other Names: FARXIGA

SUMMARY:
Cystinuria is an inherited autosomal recessive disorder of the kidney that is the result of an inability to reabsorb dibasic amino acids, including cystine, from the urine. Supersaturation of cystine in the urine produces crystals that precipitate and form stones in the kidney, which can be a cause of obstruction, infection, and chronic kidney disease. Cystine stones constitute a major health challenge for affected individuals with cystinuria because of the frequent recurrence of painful symptoms and the current absence of effective, patient-accepting treatment.

A mainstay of therapy is breaking or preventing the cystine bond on the molecular level such that cystine (which is formed from the joining of two cysteine amino acids and their corresponding sulfur atoms) cannot precipitate in the urine. It is hypothesized that a glucose molecule may be able to do this if introduced into the urine. SGLT-2 inhibitors are a class of drug that are FDA approved to treat diabetes mellitus (DM) and heart failure by inhibiting an enzyme in the kidney that allows for reabsorption of glucose from the urine. This effectively increases the concentration of glucose in the urine. The hypothesis suggests that administration of this drug to patients with cystinuria will introduce sufficient glucose into the urine to prevent or reverse the formation of cystine stones. To date, there has been no published data on the effectiveness of this therapy for this indication, although the dosage and administration would be identical to that already approved by the FDA for the treatment of DM and heart failure.

DETAILED DESCRIPTION:
This is a single center, prospective cohort trial designed to assess the effect of daily oral administration of dapagliflozin 10 mg on cystine stone formation across routine imaging obtained during management of this disease. 25 subjects are planned, each with previously diagnosed cystinuria and without current treatment except with potassium citrate medication.

Each patient identified in the clinic as a potential participant will be screened to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be entered into the study. Consent will be obtained. The therapy under investigation, dapagliflozin 10 mg, will then be administered orally to each participant daily for one year. Each subject will be contacted 1 week by the study team after treatment begins to check compliance, tolerability, and side effects with SGLT-2 inhibitor therapy. Each subject will then be contacted every 8 weeks by the study team for follow-up and to continue checks on compliance, tolerability, and side effects with SGLT-2 inhibitor therapy. Each subject will subsequently undergo routine care with no further alterations or interruptions to their typical care with routine follow up appointments with a study doctor every 3-4 months.

Routine standard-of-care surveillance imaging for their cystinuria and formation of cystine stones will also occur as part of the treatment and management of each participant's kidney stone disease. This routine care will continue to be performed during the study period, the only difference being the collection of data with regard to ongoing stone burden for the cystinuria patients receiving treatment with daily oral dapagliflozin 10 mg on each routine imaging scan. Tolerability of the study therapy will be assessed at each routine visit during the participant's usual care. Participants who require operative intervention for their kidney stones during the treatment period will be removed from the study. No placebo will be used during this study.

Total duration of subject participation with be up to 1 year and 3 months. Total duration of the study is expected to be up to 1 year and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* males and females age 18 or older
* documented cystinuria on prior 24-hour urine collection and/or stone analysis
* history of previous cystine kidney stones
* able and willing to provide consent

Exclusion Criteria:

* prior diagnosis of diabetes mellitus (type I or type II)
* vulnerable populations including incarceration status
* anticipation of pregnancy during the study duration
* unable to give informed consent
* non-English primary language
* pregnancy, lactation, or child- bearing age without birth control devices
* serious illness likely to cause death within the next 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in cystine stone size over time (1 year and 3 months) | 1 year and 3 months
  The change in cystine stone size in mm will be measured over time using routine, standard-of-care imaging obtained during the management of patients with cystinuria.

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Stoller, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No